CLINICAL TRIAL: NCT00264953
Title: HD11 for Intermediate Stages
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: German Hodgkin Study Group
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HD11
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-07

CONDITIONS: Hodgkin´s Lymphoma
Keywords: Hodgkin´s lymphoma; intermediate stages
MeSH Terms: interventions — Doxorubicin; Bleomycin; Vinblastine; Dacarbazine; Etoposide; Procarbazine; Prednisone; Vincristine; Radiotherapy

ARMS (4):
- A (Active Comparator): 4x ABVD plus 30Gy IF-RT
  Interventions: Drug: Adriamycin; Drug: Bleomycin; Drug: Vinblastine; Drug: DTIC; Radiation: radiation therapy
- C (Experimental): 4x BEACOPP baseline plus 30Gy IF-RT
  Interventions: Drug: Adriamycin; Drug: Bleomycin; Drug: Etoposide; Drug: Procarbazine; Drug: Prednisone; Drug: Vincristine; Radiation: radiation therapy
- B (Experimental): 4x ABVD plus 20Gy IF-RT
  Interventions: Drug: Adriamycin; Drug: Bleomycin; Drug: Vinblastine; Drug: DTIC; Radiation: radiation therapy
- D (Experimental): 4x BEACOPP baseline plus 20Gy IF-RT
  Interventions: Drug: Adriamycin; Drug: Bleomycin; Drug: Etoposide; Drug: Procarbazine; Drug: Prednisone; Drug: Vincristine; Radiation: radiation therapy

INTERVENTIONS:
Drug: Adriamycin
Drug: Bleomycin
Drug: Vinblastine
  Arms: A; B
Drug: DTIC
  Arms: A; B
Drug: Etoposide
  Arms: C; D
Drug: Procarbazine
  Arms: C; D
Drug: Prednisone
  Arms: C; D
Drug: Vincristine
  Arms: C; D
Radiation: radiation therapy — 20 or 30Gy IF-RT

SUMMARY:
This study is designed to (1) compare the efficacy of the BEACOPP regimen with that of ABVD as a 4-cycle chemotherapy combined with an involved field irradiation and (2) to define the optimum radiation dose comparing of 30 to 20 Gy in the same context.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin´s lymphoma (histologically proven)
* CS (PS) IA, IB, IIA, with one of the risk factors a-d CS (PS) IIB only with risk factor c or d

  1. bulky mediastinal mass (> 1/3 maximum transverse thorax diameter)
  2. extranodal involvement
  3. ESR > 50 (A), > 30 (B-symptoms)
  4. 3 or more lymph node areas involved
* written informaed consent

Exclusion Criteria:

* Leukocytes <3000/microl
* Platelets <100000/microl
* Hodgkin´s Disease as "composite lymphoma"
* Activity index (WHO) < grade 2

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1395 (Actual)
Dates: Start 1998-05; Primary Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volker Diehl, Prof., Principal Investigator — University of Cologne

REFERENCES:
- [Result] Eich HT, Diehl V, Gorgen H, Pabst T, Markova J, Debus J, Ho A, Dorken B, Rank A, Grosu AL, Wiegel T, Karstens JH, Greil R, Willich N, Schmidberger H, Dohner H, Borchmann P, Muller-Hermelink HK, Muller RP, Engert A. Intensified chemotherapy and dose-reduced involved-field radiotherapy in patients with early unfavorable Hodgkin's lymphoma: final analysis of the German Hodgkin Study Group HD11 trial. J Clin Oncol. 2010 Sep 20;28(27):4199-206. doi: 10.1200/JCO.2010.29.8018. Epub 2010 Aug 16. PMID 20713848
- [Derived] Hay AE, Klimm B, Chen BE, Goergen H, Shepherd LE, Fuchs M, Gospodarowicz MK, Borchmann P, Connors JM, Markova J, Crump M, Lohri A, Winter JN, Dorken B, Pearcey RG, Diehl V, Horning SJ, Eich HT, Engert A, Meyer RM; Conducted by the NCIC Clinical Trials Group (Canada) and German Hodgkin Study Group (GHSG). An individual patient-data comparison of combined modality therapy and ABVD alone for patients with limited-stage Hodgkin lymphoma. Ann Oncol. 2013 Dec;24(12):3065-9. doi: 10.1093/annonc/mdt389. Epub 2013 Oct 11. PMID 24121121
- [Derived] Boll B, Gorgen H, Fuchs M, Pluetschow A, Eich HT, Bargetzi MJ, Weidmann E, Junghanss C, Greil R, Scherpe A, Schmalz O, Eichenauer DA, von Tresckow B, Rothe A, Diehl V, Engert A, Borchmann P. ABVD in older patients with early-stage Hodgkin lymphoma treated within the German Hodgkin Study Group HD10 and HD11 trials. J Clin Oncol. 2013 Apr 20;31(12):1522-9. doi: 10.1200/JCO.2012.45.4181. Epub 2013 Mar 18. PMID 23509310
- See also: Description od study in German (Website of the Competence Network Malignant Lymphoma) — http://www.lymphome.de/Gruppen/GHSG/